CLINICAL TRIAL: NCT05049070
Title: A Prospective, Multicenter, Open Label Study to Evaluate the Reliability, Validity and Safety of Subjective Mobile Refraction Assessed by GoEyes
Brief Title: Study to Evaluate the Reliability, Validity and Safety of Subjective Mobile Refraction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: 1800 Contacts, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: QAD-079
Record Dates: First submitted 2021-08-23; First posted 2021-09-17 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Refractive Errors
Keywords: Refractive Errors; Myopia; Mobile Applications
MeSH Terms: conditions — Refractive Errors; Myopia

STUDY DESIGN:
Masking Description: The Best Corrected Visual Acuity (BCVA) assessor will be masked to GoEyes and Standard of Care refraction results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- GoEyes (Experimental): GoEyes Self administered refraction test + Standard of care refraction test
  Interventions: Diagnostic Test: Mobile medical application to self administer a subjective refraction test; Diagnostic Test: Standard of care refraction test

INTERVENTIONS:
Diagnostic Test: Mobile medical application to self administer a subjective refraction test — GoEyes is a software as a medical device and mobile medical application, which is downloaded to a smartphone and is a self-administered subjective refraction test that measures the refractive error of the user's eyes in the home environment without any contact or help from health care professionals
  Other Names: GoEyes
Diagnostic Test: Standard of care refraction test — Standard of care subjective manifest refraction test performed by a healthcare professional

SUMMARY:
This study evaluates the reliability, validity and safety of a self administered, subjective refraction test via a mobile medical app (GoEyes) as compared to standard of care subjective manifest refraction performed by a health care provider, in subjects who have no known ocular disease or condition other than refractive error.

DETAILED DESCRIPTION:
GoEyes is a Mobile Medical Application, which can be downloaded to a smartphone and is being developed as a self -administered subjective refraction examination that measures the refractive error of the user's eyes in the home environment without any contact or help from health care professionals.

The Study will be conducted in 2 parts; Part 1 and Part 2.

Approximately 59 participants will be enrolled In Part 1. Part 1 participants will have a GoEyes refraction test in clinic on two separate days and will also have a standard of care refraction test performed by a health care provider and best corrected visual acuity assessments.

Approximately 349 participants will be enrolled in Part 2. Part 2 participants will self administer the GoEyes test at home on 2 separate days and will also have in clinic standard of care refraction test performed by a health care provider and best corrected visual acuity assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged 18-39 years who currently wear glasses and/or soft contact lenses to correct refractive error
2. Normal color vision
3. Able to use both hands at the same time and to hear, understand and verbally respond to audio instructions
4. Have single vision lenses only
5. Able to provide informed consent -

Exclusion Criteria:

1. Have any ongoing disease or ocular condition other than refractive error
2. Have a history of permanent vison loss
3. Have a neurological condition affecting vision
4. Have worn glasses since age 6 or younger
5. Have a prism in their prescription
6. Use Rigid gas permeable lenses or OrthoK lenses
7. Have had laser refractive surgery or any other eye surgery
8. Use prescription eye drops -

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 349 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
90% Concordance for sphere power and cylinder power (monocular) | Baseline
Descriptive statistics for concordance of cylinder axis (monocular) stratified by cylinder power | Baseline
Monocular refractive outcomes | Baseline
  Lower confidence limit of ≥ 90% for concordance (for right and left eyes separately)
Monocular visual acuity | Baseline
  Lower confidence limit of ≥95% (for right and left eyes combined)
Proportion of out-of-range eye that are correctly excluded | Baseline
Incidence of Adverse Events in Part 1 | 21 days
Incidence of Adverse Events in Part 2 | 8 Days

SECONDARY OUTCOMES:
Descriptive statistics for sphere power and cylinder power (monocular) | Baseline and Visit 2 (day 2-21 for part 1 and day 2-8 for part 2)
Descriptive statistics for cylinder axis (monocular) stratified by cylinder power | Baseline and Visit 2 (day 2-21 for part 1 and day 2-8 for part 2)
Descriptive statistics for concordance of monocular refractive outcomes (for right and left eyes separately | Baseline and Visit 2 (day 2-21 for part 1 and day 2-8 for part 2)
Descriptive statistics for monocular and binocular visual acuity (for right and left eyes combined | Baseline
Proportion of out of range eyes that are correctly excluded | Baseline and Visit 2 (day 2-21 for part 1 and day 2-8 for part 2)
Comparison of test and re-test measurements to Standard of Care (SOC) data | Baseline and Visit 2 (day 2-21 for part 1 and day 2-8 for part 2)
Rate of disagreement between GoEyes screening at home and in-clinic screening | Baseline

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Matrix Clinical Research, Beverly Hills, California
  - North Bay Eye Associates, Petaluma, California
  - Empire Clinical Research, Pomona, California
  - Segal Drug Trials, Delray Beach, Florida
  - Butchertown Clinical Trials, Louisville, Kentucky
  - Tauber Eye Center, Kansas City, Missouri
  - IMA Research, Las Vegas, Nevada
  - Core, Inc Vita Eye Clinic, Shelby, North Carolina
  - Athens Eye Care, Athens, Ohio
  - Optimed Research, Marysville, Ohio
  - Total Eye Care, Memphis, Tennessee
  - Wagner Macula & Retina, Norfolk, Virginia